CLINICAL TRIAL: NCT04940351
Title: Comparative Evaluation of the Effectiveness of Piezocision and Micro-osteoperforation in Alleviating Mandibular Anterior Crowding: A Randomized Clinical Trial
Brief Title: Evaluation of the Effectiveness of Piezocision and Micro-osteoperforation in Alleviating Mandibular Anterior Crowding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANANDA RAJ S PGIDS/BHRC/21/19
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Crowding of Anterior Mandibular Teeth
Keywords: dental crowding
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP - A: PIEZOCISION GROUP (Experimental): This group will receive piezocision using piezotome inbetween the roots of mandibular anteriors after the placement of initial arch wire.
  Interventions: Procedure: GROUP - A: PIEZOCISION GROUP
- GROUP- B: MICRO-OSTEOPERFORATION GROUP (Experimental): This group will receive Micro-Osteoperforation using orthodontic mini-implants and mini-implant screw driver after the placement of initial arch wire.
  Interventions: Procedure: GROUP- B: MICRO-OSTEOPERFORATION GROUP

INTERVENTIONS:
Procedure: GROUP - A: PIEZOCISION GROUP — This group will receive piezocisions after placement of initial arch wire, in between the roots of mandibular anteriors (in a vertical line) i.e., between mandibular canine and lateral incisors bilaterally, lateral incisors and central incisors bilaterally and between two cental incisors with the help of piezotome. These piezocisions will be performed on the labial cortical bone only, 4mm below the interdental papilla under 2% lidocaine with 1:100,000 epinephrine and with standard asepsis, and gingival overlying will be incised first with blade number 15 in a Bard Parker handle. A piezosurgical microsaw with piezosurgical drill will be placed over that incision with irrigation. Then, vertical 5- to 8-mm and 3mm deep corticotomies will be perform using periapical radiographs as a guide to avoid penetrating into the adjacent roots. No subsequent sutures required.
  Arms: GROUP - A: PIEZOCISION GROUP
Procedure: GROUP- B: MICRO-OSTEOPERFORATION GROUP — This group will receive MOPs after initial arch wire placement. These MOPs will be performed under local anesthesia with standard asepsis, using a self drilling 1.6mm x 8mm orthodontic mini-implants and mini-implant screw driver and no flap will be raised. MOP's will be placed on five sites i.e., interproximally between mandibular canine and lateral incisors bilaterally, central incisor and lateral incisor bilaterally and between two central incisors. Each site will receive two MOP's, first 2mm apical to alveolar crest and second 2mm below the first in a vertical line and 2mm deep into the bone. Then the mini-implant will be removed by rotating the screw driver anticlockwise and pressure will be applied to achieve hemostasis.
  Arms: GROUP- B: MICRO-OSTEOPERFORATION GROUP

SUMMARY:
In recent times, many patients want their treatment duration to be reduced, because lengthy orthodontic treatment duration is associated with negative sequelae such as discomfort, pain, white spot lesions, and decreased patient's compliance. Several techniques have been employed in an attempt to accelerate the tooth movement and shorten the lengthy orthodontic treatment duration. So, this study will investigate the effectiveness of minimal invasive technique like piezocision and microosteoperforation in alleviating mandibular anterior crowding which is one of the common malocclusiom and provide scientific knowledge regarding which minimal invasive tecnique will relieve the crowding faster.

DETAILED DESCRIPTION:
Records will be taken from patients who are meeting selection criteria and then analysis of record will be done to attain a proper diagnosis and treatment plan. Afterthat, those patients will be referred to oral surgery department for extraction of first premolar. After healing, orthodontic treatment will be started with bonding of preadjusted MBT 0.022" slot straight wire appliance(Patient will be instructed to report immediately in case of breakage of appliance), after that, randomisation and allocation of two groups will be done and on the day of initial aligning archwire placement i.e., 0.014" NiTi, active interventions(piezocision and micro-osteoperforations) will be done for each group and then levelling and alignment will be continued with the following arch wire sequence 0.016" , 0.016" x 0.022" and 0.017" x 0.025" NiTi. Levelling and alignment will be considered finished when 0.017x0.025" NiTi archwire will be engaged passively in the brackets. Records i.e,. mandibular study models will be taken on the day of surgical procedure before surgery (T0) and then after every 4th week i.e., 4th week(T1), 8th week(T2), 12th week(T3), 16th week(T4). Following this, data collection and interpretation of results will be done. And also, CBCT will be taken at post levelling and alignment with 0.017" x 0.025" arch wire to assess the root resorption and marginal alveolar bone loss.

ELIGIBILITY:
Inclusion Criteria:

Patient satisfying the following criteria will be included in this clinical study:

1. Patients with age between 16-25 years
2. Patients with either Angle's class I or class II malocclusion with moderate crowding in the anterior mandible(LII- 4-6mm) who requires extraction in the lower arch (tooth-size-arch-length discrepancy>5 mm)
3. Permanent dentition
4. Existence of all tooth in the mandibular arch (except third molars which may or may not be present)
5. Good oral hygiene and periodontal health
6. No smoking habit.

Exclusion Criteria:

1. medical conditions that would affect tooth movement (corticosteroid treatments, NSAIDs consumption, bisphosphonates, hyperparathyroidism, osteoporosis, uncontrolled diabetes)
2. Contraindication to oral surgery (medical, social, psychological)
3. Missing tooth in the mandibular arch
4. Presence of primary or supernumerary tooth in mandibular arch
5. Previous orthodontic treatment
6. Poor oral hygiene and current periodontal disease
7. Smoking habit.

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Amount of Crowding Relieved | 4 weeks
  Measured with Little Irregularity index using Digital caliper
Amount of Crowding Relieved | 8 weeks
  Measured with Little Irregularity index using Digital caliper
Amount of Crowding Relieved | 12 weeks
  Measured with Little Irregularity index using Digital caliper
Amount of Crowding Relieved | 16 weeks
  Measured with Little Irregularity index using Digital caliper

SECONDARY OUTCOMES:
Overall Alignment Time | 16 weeks
  Time taken to align the mandibular anteriors calculated in days
Root resorption of mandibular anteriors | 16 weeks
  Root length of mandibular anteriors measured before and after alignment using CBCT
Marginal Alveolar Bone Loss | 16 weeks
  Alveolar bone length measured before and after alignment using CBCT

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No